CLINICAL TRIAL: NCT03243435
Title: Feasibility of Breast MRI After Sentinel Procedure for Breast Cancer With Superparamagnetic Tracers
Brief Title: Sienna+MR Long-term Uptake
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Cornelia Leo, Head, Breast Center, Kantonsspital Baden
Other Study IDs: 2016-00808
Record Dates: First submitted 2016-07-05; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Native 1,5 Tesla breast MRI group: From all patients a 1,5 Tesla MRI of the breast will be obtained
  Interventions: Procedure: Native 1,5 Tesla breast MRI

INTERVENTIONS:
Procedure: Native 1,5 Tesla breast MRI

SUMMARY:
In a previous study in 2012/2013 patients were injected a superparamagnetic iron oxide for sentinel lymph node detection. In this follow up study we want to investigate how much of this tracer is still detectable.

ELIGIBILITY:
inclusion:

* participation in previous study
* informed consent
* no contraindications for MRI scan

exclusion:

* contraindications for MRI scan

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all 34 patients from the previous study are included
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
I) Analysis if the supraparamegnetic Tracer is still detectable | 04/2017
  Analysis by two expert radiologists

SECONDARY OUTCOMES:
Analysis to which degree of impairment of Imaging is detected | 04/2017
  Description as "no impairment", impairment, but Interpretation of Images possible", "impairment, Image Interpretation impossible"

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No